CLINICAL TRIAL: NCT02421133
Title: Impact of a Transitional Care Program Involving an Advanced Practice Nurse on 30-Day Hospital Readmissions for Elderly Patients Discharged From a Short Stay Geriatric Ward (PROUST Study)
Brief Title: Impact of a Transitional Care Program on 30-Day Hospital Readmissions for Elderly Patients Discharged From a Short Stay Geriatric Ward
Acronym: PROUST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2014.874
Record Dates: First submitted 2015-03-09; First posted 2015-04-20 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Geriatrics
Keywords: Care transition program; Patient readmission; Transition Nurse; Stepped wedge; elderly

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transitional care program. (Experimental): The transitional care program from hospital to home will be implemented at three steps: during the patient's stay in hospital, the day of the discharge and during 4 weeks after discharge.
  Interventions: Other: Transitional care program.
- standard care program (Other): No intervention liable to affect the care provided to the patients, the organization of care or the practices of health care professionals will be implemented during the control period (time steps without intervention).
  Interventions: Other: standard care program

INTERVENTIONS:
Other: Transitional care program. — During the patient's stay in hospital, the transition nurse creates a transitional care file including information about the patient (inpatient medical and nurse care plan, medications), the discharge plan, and the contact information of the relevant primary care providers. She notifies the patient's primary care physician of the date of the discharge to home, of the potential medical problems and of the discharge care plan; a primary care physician visit is planned the month following the discharge.
  The day of the hospital discharge: meeting with the patient to review the follow-up recommendations. The transition nurse verifies that the medications are prescribed accordingly with the discharge plan, that the patient and his caregiver understand the prescription and are informed with the planned appointments and the biological monitoring.
  During 4 weeks after the hospital discharge: follow-up by the transition nurse once a week, alternately by telephone and home visit.
  Arms: Transitional care program.
Other: standard care program — The patients will be discharged according to the usual care plan of each participating hospital. The medical team does a medical and geriatric assessment of the patients according to the recommendations. The communication of information to the primary care providers (nurse, primary care physician…) is left to the discretion of the medical teams of the discharging hospitals, according to their habits of work.
  Arms: standard care program

SUMMARY:
In France, it has be estimated that the hospital readmission rate within 30 days of patients aged 75 or older is 14% (IC95% [12.0-16.7]), nearly a quarter being avoidable. There is evidence that interventions "bridging" the transition from hospital to home involving a dedicated professional (usually nurses) would be most effective in reducing the risk of readmission, but the level of evidence of current studies is low. Our study aims to assess the impact of a program of transitional care from hospital to home for people of 75 years old or more admitted to acute care.

DETAILED DESCRIPTION:
The study is a stepped wedge randomized cluster study. Intervention: The transition care program, involving a dedicated advanced practice nurse, will include: 1) during the patient's stay in hospital: an individualized needs-based comprehensive discharge plan and a transitional care record ; the notification of the primary care physician about inpatient care and hospital discharge; 2) the day of the discharge: specific explanations about the organization of home care provided by the transition care nurse to the patient; 3) during 4 weeks after discharge: monitoring patients and caregivers regularly through home visits and/or telephone contact,

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized for 48 hours or more in one of the acute geriatric service participating to the study.
* Aged 75 or older.
* Leaving at home and with home as the planned discharge after the admission.
* At risk of hospital readmission emergency visit rates after discharge (if he has two or more of the following criteria (taken from the Triage Risk Screening Tool and from the 2013 French recommendation)).

Exclusion Criteria:

* Patient leaving in a retirement home.
* Patient hospitalized at home.
* Patient leaving at home but at 30 km (18 miles) or more from the service of his index admission

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 630 (Actual)
Dates: Start 2015-07; Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
30-Day unscheduled hospital readmission or emergency visit rate after the index hospital discharge. | Within 30 days after hospital discharge.
  Unscheduled hospital readmissions are hospitalizations that are not planned at the moment of the discharge (for example: hospitalization after an emergency visit or upon request of the primary care physician).

SECONDARY OUTCOMES:
Length of stay in the short stay geriatric ward (index hospitalization) | Patients will be followed for the duration of hospital stay, an expected average between 2 days and 30 days
Unscheduled hospital readmissions or emergency room visits | Within 30 and 90 days after the index hospital discharge.
Free-hospitalization survival | Within 30 and 90 days after the index hospital discharge.
Mortality rate | Within 30 and 90 days after the index hospital discharge.
Adverse events (i.e. falls) | Within 30 days after the index hospital discharge.
Quality of life. | Within 30 days after the index hospital discharge.
  Measured with the French version of the EUROQOL-5D.
Patients' satisfaction care transition programme | Within 30 days after the index hospital discharge.
  Measured with the Care Transition Measure® questionnaire.
Delay between the index hospital discharge and the implementation of home care. | Within 30 days after the index hospital discharge.
Number of contacts between the transition nurse and the primary care providers or the hospital providers after discharge | Within 30 days after the index hospital discharge.
Costs of unscheduled hospital readmission or emergency visit | 30 days after discharge
  Hospital and community care costs after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Marc Bonnefoy, Principal Investigator — Centre Hospitalier Lyon Sud-Hospices Civils de Lyon
Locations (9):
- France (9):
  - CH Gériatrique des Monts d'Or, Albigny-sur-Saône
  - CH Bourg-en-Bresse, Bourg-en-Bresse
  - Centre Hospitalier Alpes Léman, Contamine-sur-Arve
  - Hôpital Édouard Herriot, Lyon
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHG Annecy, Pringy
  - CH Saint-Chamond, Saint-Chamond
  - Clinique des portes du sud, Vénissieux
  - CH Villefranche, Villefranche

REFERENCES:
- [Result] Occelli P, Touzet S, Rabilloud M, Ganne C, Poupon Bourdy S, Galamand B, Debray M, Dartiguepeyrou A, Chuzeville M, Comte B, Turkie B, Tardy M, Luiggi JS, Jacquet-Francillon T, Gilbert T, Bonnefoy M. Impact of a transition nurse program on the prevention of thirty-day hospital readmissions of elderly patients discharged from short-stay units: study protocol of the PROUST stepped-wedge cluster randomised trial. BMC Geriatr. 2016 Mar 3;16:57. doi: 10.1186/s12877-016-0233-2. PMID 26940678